CLINICAL TRIAL: NCT06064747
Title: Low-Frequency REpetitive TRanscranial Magnetic Stimulation Combined With Endovascular Treatment in ACute Ischemic StrokE (RETRACE-II): A Randomized, Double-Blind, Sham-Controlled, Phase 2 Pilot Trial
Brief Title: Low-Frequency REpetitive TRanscranial Magnetic Stimulation Combined With Endovascular Treatment in ACute Ischemic StrokE
Acronym: RETRACE-II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yongjun Wang, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HX-A-2023002
Record Dates: First submitted 2023-08-24; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Stroke, Acute Ischemic
Keywords: Acute ischemic stroke; LF-rTMS; Endovascular therapy; Phase 2 Pilot Trial
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: In order to ensure the blind method, the sham stimulation coil was used, which had the same parameters (including location, stimulation frequency, time, etc.) as the LF-rTMS group, and had the same stimulation sound to ensure no effective stimulation, to ensure the blind state is maintained during the test. Investigators and patients who participated in the study treatment or involved in the clinical evaluation of patients were blinded to treatment grouping.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LF-rTMS (Experimental): Using "8" coil,1-Hz rTMS to stimulate the M1 region of the ipsilateral hemisphere, the stimulation intensity was RMT 100%, 1200pulses/session, two sessions (2400 pulses)/day (interval ≥ 2 hours), lasting 3 days (total 6 sessions, 7200pulses)
  Interventions: Device: LF-rTMS
- Sham coil stimulation (Sham Comparator): The sham stimulation coil was used to stimulate the same site, duration and sound as the LF-rTMS group, ensuring no effective stimulation, twice a day for 3 days
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: LF-rTMS — LF-rTMS group: using "8" coil,1-Hz rTMS to stimulate the M1 region of the ipsilateral hemisphere, the stimulation intensity was RMT 100%, 1200pulses/session, two sessions (2400 pulses)/day (interval ≥ 2 hours), lasting 3 days (total 6 sessions, 7200pulses);
  Arms: LF-rTMS
Device: Sham stimulation — Sham stimulation group: the sham stimulation coil was used to stimulate the same site, duration and sound as the LF-rTMS group, ensuring no effective stimulation, twice a day for 3 days.
  Arms: Sham coil stimulation

SUMMARY:
This is a multicenter, randomized, double-blind, sham-controlled, investigator-initiated clinical study, to evaluate the clinical efficacy and safety of LF-rTMS in rescuing the ischemic penumbra, reducing disability rate and improving functional outcome in patients with acute ischemic stroke receiving early endovascular recanalization (bridging or direct endovascular therapy)

DETAILED DESCRIPTION:
The target population of this study was patients with acute ischemic stroke of the anterior circulation diagnosed clinically. The site of acute occlusion of the responsible vessel was located in the intracranial segment of the internal carotid artery, T-type bifurcation or M1 segment of the middle cerebral artery, planning for bridging therapy (bridging intravascular therapy after intravenous thrombolysis with alteplase) or direct intravascular therapy, the time from stroke onset to the start of the trial intervention was less than 24 hours (when the exact time of onset was unknown, the patient's"Last apparent normal time" was defined as the time of onset).

Enrolled patients were randomly assigned in a 1:1 ratio to the"LF-rTMS group" or the"Sham Stimulation Group" and received:

1. LF-rTMS group: using "8" coil,1-Hz rTMS to stimulate the M1 region of the ipsilateral hemisphere, the stimulation intensity was RMT 100%, 1200pulses/session, two sessions (2400 pulses)/day (interval ≥ 2 hours), lasting 3 days (total 6 sessions, 7200pulses);
2. Sham stimulation group: the sham stimulation coil was used to stimulate the same site, duration and sound as the LF-rTMS group, ensuring no effective stimulation, twice a day for 3 days.

All patients received endovascular therapy (bridging therapy or direct endovascular therapy).

All patients were followed up until the 90th day after randomization to evaluate the clinical efficacy and safety of LF-rTMS in rescuing the ischemic penumbra, reducing disability rate and improving functional outcome in patients with acute ischemic stroke receiving early endovascular recanalization (bridging or direct endovascular therapy)

ELIGIBILITY:
Inclusion Criteria:

1. 18 - 80 years, male or female;
2. Clinically diagnosed as acute anterior ischemic stroke, artery occlusion occurred at the terminal of the intracranial carotid artery, T-shaped bifurcation or M1 segment of the middle cerebral artery;
3. Within 24 hours of stroke onset;
4. Eligible for other imaging indications for bridging therapy or direct mechanical thrombectomy:

   ASPECTS ≥6 certified by the latest brain CT imaging; Patients within 6-16 hours after stroke onset should meet the mismatch criteria, which was defined as infarction core volume <70 ml, mismatch ratio ≥1.8 and the ischemic volume > 15 ml (DEFUSE-3 Criteria); or NIHSS score ≥ 10 with infarction -core volume < 31 cm3, or NIHSS score ≥ 20 with infarction core volume ≤ 51 cm3 (DAWN Criteria); Patients within 16-24 hours after stroke onset should meet the mismatch criteria, which was defined as NIHSS score ≥ 10 with infarction-core volume < 31 cm3, or NIHSS score ≥ 20 with infarction-core volume ≤ 51 cm3 (DAWN Criteria);
5. Planned to receive bridging therapy (endovascular therapy after intravenous alteplase) or direct endovascular therapy;
6. Pre-morbid modified Rankin Scale ≤1;
7. 6 ≤ NIHSS ≤ 25 before endovascular therapy;
8. Signed informed consent from subjects or legally authorized representatives

Exclusion Criteria:

1. TMS contraindications include metallic foreign bodies in the head, pacemaker, implantable drug pumps, cochlear implants, etc.
2. Epilepsy or history of epilepsy, intracranial hypertension, tumor and other serious neurological disorders;
3. Midline displacement and brain parenchymal mass effect seen in head CT and other images;
4. Head CT or MRI showed bilateral acute cerebral infarction;
5. CT or MRI showed a large area of infarction (> 1/3 of the area supplied by middle cerebral artery);
6. Evidence of acute intracranial hemorrhage;
7. Before the bridging therapy, other thrombolytic drugs besides alteplase or tenecteplase were used;
8. A history of congenital or acquired hemorrhagic disease, coagulation factor deficiency, or thrombocytopenia disease;
9. After blood pressure control, the systolic blood pressure was still ≥180 mmHg or the diastolic blood pressure was ≥110 mmHg;
10. Known recent or current serum creatinine exceeding 1.5 times the upper limit of normal or estimated glomerular filtration rate (EGFR) < 60 mL/min;
11. Patients during pregnancy or lactation and within 90 days of planned pregnancy;
12. Patients with severe mental disorders or dementia who can not cooperate with informed consent and follow-up;
13. Patients with malignancy or severe systemic disease and expected survival of less than 90 days;
14. Participants in other clinical intervention studies within 30 days before randomization or who were participating in other clinical intervention studies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-08 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Rescue penumbra ratio | 3 days
  Baseline penumbra volume - Infarct volume 3 days after randomization / Baseline penumbra volume × 100%
Early neurological improvement (ENI) | 3 days
  The proportion of patients with a reduction of ≥4 on the NIHSS, compared with the baseline score or an NIHSS of 0 or 1
Symptomatic intracranial hemorrhage | 3 days
  The proportion of symptomatic intracranial hemorrhage

SECONDARY OUTCOMES:
Infarct volume progression | 3 days
  The difference between CT infarct volume and baseline core infarct volume
Final infarct volume | 7 and 90 days
  Infarct volume on DWI at day 7 after randomization, and infarct volume on FlAIR at Day 90 ± 7 after randomization.
mRS scores of 0-1 | 90 days
  Proportion of patients with mRS scores of 0-1
mRS scores of 0-2 | 90 days
  Proportion of patients with mRS scores of 0-2
Secondary brain injury on imaging | 90 days
  Evaluation of cerebral infarction volume on FLAIR and cerebral atrophy
Barthel index of ADL | 90 days
  Barthel index of ADL, 0-100 (higher score indicates better)
EQ-5D-5L | 90 days
  The Health Questionnaire (EQ-5D-5L) is a self-report survey that measures quality of life across 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is scored on a 5-level severity ranking that ranges from "no problems" through "extreme problems."
Montreal Cognitive Assessment (MoCA) total score | 90 days
  Total score of the MoCA Performance on the MoCA (0-30; higher score indicates better performance)
Serious adverse events (SAE) | 90 days
  The proportion of serious adverse events (SAE)
All-cause deaths | 90 days
  The proportion of all-cause deaths
Symptomatic intracranial hemorrhage | 90 days
  The incidence of symptomatic intracranial hemorrhage
Deterioration of neurological function | 3 days
  The incidence of deterioration of neurological function (NIHSS increase ≥4 points)
Stroke recurrence | 90 days
  Cerebral infarction, cerebral hemorrhage
Adverse events (AE) | 3 days
  Adverse events (AE)

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun MD Wang, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tian tan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ding L, Wang W, Yi T, Zhang G, Han X, Chen W, Wang H, Wang Y, Li Z. Rationale and design of Low-Frequency REpetitive TRanscranial Magnetic Stimulation Combined with Endovascular Treatment in ACute Ischaemic StrokE (RETRACE II): a randomised double-blind controlled multicentre phase II pilot study. Stroke Vasc Neurol. 2025 Oct 28:svn-2025-004331. doi: 10.1136/svn-2025-004331. Online ahead of print. PMID 40721316